CLINICAL TRIAL: NCT02457429
Title: A Validation Study of the Dx-pH Probe in Children for the Detection of Extra-oesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01843
Record Dates: First submitted 2015-03-31; First posted 2015-05-29 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Gastro-oesophageal Reflux
Keywords: Gastro-oesophageal reflux; Children; Dx-pH Pharyngeal probe; GORD; Trans-nasal catheter
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Routine oesophageal pH monitoring (Other): Routine oesophageal pH investigation involves the trans-nasal placement of a microelectrode into the distal oesophagus as per hospital protocol. Examining the oropharynx and confirming visualisation of the red LED at the catheter tip in the correct position just below the soft palate will confirm its position in the oropharynx. The internal pH value of the oesophagus is then continuously measured and recorded onto a small ambulatory device. The 2 catheters are connected to the ambulatory recording devices and recording commences. The duration of the investigation is 24 hours.
  Interventions: Device: Experiemental diagnostic procedure: Dx-pH measurement system; Other: Peptest assay; Other: GORD symptom questionnaire

INTERVENTIONS:
Device: Experiemental diagnostic procedure: Dx-pH measurement system — The Dx-pH Measurement system (Dx-pH; Respiratory Technology Corp., San Diego, CA) is a sensitive and minimally invasive transnasal device for detection of aerosolized extra-oesophageal acid reflux in the posterior oropharynx.
  The sterile single use Dx-pH catheter will be passed trans-nasally into the same nostril as the same nostril as the other catheter. The internal pH value of the oesophagus is then continuously measured and recorded onto a small ambulatory device. The 2 catheters are connected to the ambulatory recording devices and recording commences. The duration of the investigation is 24 hours.
Other: Peptest assay — A saliva sample of 0.5-1 ml will then be taken for pepsin assay (Peptest). The saliva sample will be drawn into a micro-centrifuge tube (0.5ml) and centrifuged. 80 microlitres is taken from the supernatant layer, vortex mixed, then applied to the assay test strip. The result is obtained after 15 minutes. The saliva sample will then be securely disposed.
Other: GORD symptom questionnaire — A validated 7 domain GORD symptom questionnaire (GSQ-YC) to quantify the GORD related symptoms their child suffers with is to be completed prior to any intervention.
  Other Names: (GSQ-YC)

SUMMARY:
Gastro-oesophageal reflux (GORD) and its extraoesophageal manifestations present with a variety of symptoms in both adult and paediatric populations. In children the effects of refluxate above the upper oesophageal sphincter (UES) has been implicated as a contributory factor in the underlying pathological processes of a number of conditions including apnoea, asthma, chronic cough, subglottic stenosis, chronic rhinosinusitis and otitis media. The absence of typical symptoms in addition to the inability to obtain a formal symptom history from a young paediatric population contributes to the difficulty in establishing a diagnosis. At present there are no studies or data directly measuring extraoesophageal reflux and its correlation to oesophageal pH monitoring in children.

The use of twenty-four hour oesophageal pH monitoring is regarded as the established technique for diagnosis of GORD, however this technique has been less reliable for detecting extra-oesophageal reflux. The investigators intend to use the Dx-pH Measurement system, a sensitive and minimally invasive transnasal device, to assess the feasibility and validate its use in a paediatric population.

DETAILED DESCRIPTION:
Gastro-oesophageal reflux (GORD) and its extraoesophageal manifestations present with a variety of symptoms in both adult and paediatric populations. In children the effects of refluxate above the upper oesophageal sphincter (UES) has been implicated as a contributory factor in the underlying pathological processes of a number of conditions including apnoea, asthma, chronic cough, subglottic stenosis, chronic rhinosinusitis and otitis media.

The absence of typical symptoms in addition to the inability to obtain a formal symptom history from a young paediatric population contributes to the difficulty in establishing a diagnosis.

At present there are no studies or data directly measuring extraoesophageal reflux and its correlation to oesophageal pH monitoring in children. As a result there is no baseline data for a paediatric population and subsequently no measureable definition of a significant extraoesophageal reflux event. There is a poor correlation between reflux events measured with an oesophageal probe and extra-oesophageal symptoms of reflux. Studies have demonstrated that 51% of patients without pharyngeal reflux had abnormal distal oesophageal pH studies.

This is secondary to both technical concerns regarding the ability of such probes in detecting aerosolized and vapour forms of reflux in the pharynx and due to the inadequacy of the definition of a significant reflux event above the upper oesophageal sphincter. Moving cephaled (upwards) within the upper aerodigestive tract will result in shorter, higher pH events that may not be recognised using traditional oesophageal analysis, which define a pH<4 as defining a significant oesophageal reflux event.

The use of twenty-four hour oesophageal pH monitoring is regarded as the established technique for diagnosis of GORD, however this technique has been less reliable for detecting extra-oesophageal reflux.

The Dx-pH Measurement system (Dx-pH; Respiratory Technology Corp., San Diego, CA) is a sensitive and minimally invasive transnasal device for detection of aerosolized extra-oesophageal acid reflux in the posterior oropharynx.

The investigators intend to use the Dx-pH measurement system and the Peptest salivary pepsin assay (RBiomed, UK) in children already undergoing oesophageal pH studies. The investigators aim to assess the feasibility of these systems in a paediatric population,to provide baseline data and to validate its use in measuring extra-oesophageal reflux events in children. These results will be correlated against symptom questionnaire scores and the results of the 24 hour oesophageal pH study results.

The investigators' results will guide further interventional studies in this area, with the eventual aim of improving diagnosis and guided treatment for the extra-oesophageal manifestations of GORD

ELIGIBILITY:
Inclusion Criteria:

* All children between the age of 1 year old and 16 years old consecutively referred for outpatient 24 hour oesophageal pH / impedance monitoring will be invited to participate in the study. This is regardless of the underlying diagnosis, aetiology and manifestation of symptoms.

Exclusion Criteria:

* Children under the age of 1 year old. Children under 1 year old will be excluded due to the technical difficulty of placing both the pH / impedance monitoring probe and the Dx-pH probe into the same nostril. Firstly, this is due to the size restriction of placing 2 probes into one nostril. Secondly, the non-pathologic high incidence of regurgitation and positing in below the age of 1 will make data difficult to interpret.
* Children with an nasogastric feeding tube in situ will be excluded. Firstly due to the difficulty in placing and securing the nasogastric, oesophageal pH and Dx-pH probe (3 tubes / probes) through the nostrils, with resultant bilateral nasal obstruction. Secondly, the nasogastric tube causes increased iatrogenic reflux within the pharynx, making data more difficult to interpret and creating artificial reflux events.
* Children with cleft palate prior to surgical repair will be excluded as the Dx-pH probe will be difficult to locate in the oropharynx and may displace into the oral cavity.
* Children requiring pH monitoring as inpatients during an acute medical admission. Children will be excluded from the study if their condition has necessitated an acute hospital admission, therefore participation in the study will not affect other ongoing investigations, treatment or their acute condition.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
pH readings from Dx-pH measurement system | 24 hours
  Baseline pH readings from Dx-pH measurement system. Measuring reflux events at pH <4, <4.5, <5.0 and <6.0.
pH readings from Dx-pH measurement system | 24 hours
  Baseline pH readings from Dx-pH measurement system. Measuring events per hour at pH <4, <4.5, <5.0 and <6.0
pH readings from Dx-pH measurement system | 24 hours
  Baseline pH readings from Dx-pH measurement system. Measuring total reflux time at pH <4, <4.5, <5.0 and <6.0.
pH readings from Dx-pH measurement system | 24 hours
  Baseline pH readings from Dx-pH measurement system. Measuring percentage reflux time at pH <4, <4.5, <5.0 and <6.0.
pH readings from Dx-pH measurement system | 24 hours
  Baseline pH readings from Dx-pH measurement system. Measuring the longest reflux period at pH <4, <4.5, <5.0 and <6.0.

SECONDARY OUTCOMES:
Conventional oesophageal pH / impedance readings | 24 hours
  Number of reflux events at pH <4, <4.5, <5.0, <6.0 will be measured.
Conventional oesophageal pH / impedance readings | 24 hours
  Number of events per hour at pH <4, <4.5, <5.0 and <6.0 will be measured.
Conventional oesophageal pH / impedance readings | 24 hours
  Total reflux time at pH <4, <4.5, <5.0, <6.0 will be measured.
Conventional oesophageal pH / impedance readings | 24 hours
  Percentage reflux time at pH <4, <4.5, <5.0, <6.0 will be measured.
Conventional oesophageal pH / impedance readings | 24 hours
  The longest reflux period. at pH <4, <4.5, <5.0, <6.0 will be measured.
GORD related symptoms (GSQ-YC) | At time of measurement
  A validated 7 domain GORD symptom questionnaire (GSQ-YC) to quantify the GORD related symptoms their child suffers with.
Pepsin (Peptest) | 15 minutes
  A saliva sample of 0.5-1ml will then be taken for pepsin assay (Peptest). The saliva sample will be drawn into a microcentrifuge tube (0.5ml) and centrifuged. 80 microlitres is taken from the supernatant layer, vortex mixed, then applied to the assay test strip.

CONTACTS AND LOCATIONS:
Overall Officials: Iain A Bruce, Principal Investigator — Royal Manchester Children's Hospital
Locations (1):
- Royal Manchester Children's Hospital, Manchester, United Kingdom